CLINICAL TRIAL: NCT05135481
Title: Effect of Intensive Lactation Support vs Frenotomy on the Incidence of Breastfeeding in Term Infants: a Randomised Control Trial
Brief Title: Dedicated Lactation Support in Infants With Tongue - Tie; a Randomised Control Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment problems
Sponsor: Princess Anna Mazowiecka Hospital, Warsaw, Poland (Other)
Collaborators: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FRENO
Record Dates: First submitted 2021-11-01; First posted 2021-11-26 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Ankyloglossia; Breast Feeding, Exclusive; Lactation Failure; Tongue-tie
MeSH Terms: conditions — Ankyloglossia; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (Active Comparator): The qualification for phrenectomy in group 1 will be made based on the Amir scale, i.e. a score of 4 and fewer points for the language function.
  Interventions: Procedure: phrenectomy
- STUDY GROUP (Experimental): Management in group 2 will include increased lactation care both during hospital stay and post discharge.
  Increased lactation care will consist of:
  individual consultations on how to properly attach the baby to the breast (at least 3 meetings during hospitalization with personnel trained in lactation counselling), regular (at least once a week) contact with a breastfeeding consultant as part of a closed group on social media or by phone, if necessary (expressed by the mother or based on a referral by a member of the lactation team) an outpatient appointment at the breastfeeding clinic.
  Interventions: Other: Increased lactation support

INTERVENTIONS:
Procedure: phrenectomy — The qualification for phrenectomy in group 1 will be made based on the Amir scale, i.e. a score of 4 and fewer points for the language function (2).
  Arms: CONTROL GROUP
Other: Increased lactation support — Management in group 2 will include increased lactation care both during hospital stay and post discharge.
  Other Names: dedicated lactation support
  Arms: STUDY GROUP

SUMMARY:
The investigators are registering a randomised controlled trial to assess whether dedicated, intensified lactation support is as good as frenotomy on the incidence of breastfeeding among term infants with ankyloglossia.

DETAILED DESCRIPTION:
The investigators plan to include a total 316 infants. The study will be carried out in level III hospital in Warsaw, Poland. The primary outcome will be exclusive breastfeeding at 12 weeks of age. Secondary outcomes include breastfeeding > 50% of feedings, improved breastfeeding comfort as assessed by the mother, weight gain, head circumference and length gain, the need to use a breast pump or lactation accessories, time of breastfeeding cessation, the type of lactation, neurological and rehabilitation assistance received, the frequency of obtained lactation, neurological and rehabilitation assistance.

ELIGIBILITY:
Inclusion criteria:

1. full - term infants born with an Apgar score of 8-10 points
2. no visual causes of lactation difficulties (malocclusion, posterior and small jaw, cervical torticollis, significant positional asymmetry)
3. parental consent

Exclusion criteria:

1. hypotrophy
2. low birth weight
3. perinatal complications
4. congenital craniofacial defects
5. neurological diseases
6. visible genetic syndromes
7. mother' unwilling to breastfeed
8. no consent for vaccination against hepatitis B
9. neonates born to HIV seropositive mothers

Ages: 1 Minute to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of exclusively breastfeeding mothers | at 12 weeks of age
  Proportion of exclusively breastfeeding mothers

SECONDARY OUTCOMES:
Proportion of mother-baby dyads with a breastfeeding frequency of > 50%. | at 12 weeks of age
  Proportion of mother-baby dyads with a breastfeeding frequency of > 50% of feedings, which will be assessed using the Breastfeeding Self-Efficacy Scale Short Form [9, 10]
Weight change | at 12 weeks of age
  Median weight change
Head circumference change | at 12 weeks of age
  Median head circumference change
Length change | at 12 weeks of age
  Median length change
Incidence of using a breast pump or lactation accessories | at 12 weeks of age
  Proportion of mothers needing to use a breast pump or lactation accessories (e.g. nipple shields)
Time of breastfeeding cessation | during 12 weeks of age
  median time of breastfeeding cessation
Rate of additional consultations | during 12 weeks of age
  Rate of consultations (e.g. speech therapist, rehabilitants, other lactation consultants) received by a mother - baby dyads.
Change in breastfeeding comfort | at 12 weeks of age
  Proportion of mothers reporting change in breastfeeding comfort

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Seliga - Siwecka, MD PhD, Study Director — Medical University of Warsaw; Justyna Fiałkowska, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of Neonatology and Neonatal Intensive Care Warsaw Medical University, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided